CLINICAL TRIAL: NCT02369068
Title: A Double-Blind, Randomized Study to Compare Onabotulinumtoxin A Versus Kenalog for Intravaginal Trigger Point Injections in the Treatment of Chronic Pelvic Pain
Brief Title: Onabotulinumtoxin A Versus Kenalog for Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamie Bartley, DO (Other)
Responsible Party: Sponsor-Investigator, Jamie Bartley, DO, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-008
Record Dates: First submitted 2015-02-05; First posted 2015-02-23 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Botulinum Toxins, Type A; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Onabotulinumtoxin A (Experimental): Intervention is a one time 30 cc intravaginal injection totaling a dose of 200u of onabotulinumtoxin A and saline injected throughout the pelvic floor at 1, 3, 5, 7, 9 and 11 o'clock sites/locations.
  An injection of 30 cc of ropivicaine (5cc/6 sites) will be used, followed by a mixture of 200 u of Onabotulinumtoxin A and 6 cc of saline (1cc/injection site).
  Interventions: Drug: Onabotulinumtoxin A
- Kenalog (Active Comparator): Intervention is a one time 30 cc intravaginal injection totaling a dose of 40mg/cc of Kenalog (triamcinolone) and ropivicaine 0.5% (29cc) injected throughout the pelvic floor at 1, 3, 5, 7, 9 and 11 o'clock sites/locations.
  A mixture of 40mg/1 cc of triamcinolone (40 mg) and 29cc of ropivicaine 0.5% (5cc/6 sites) will be used, followed by 6 cc of saline (1cc/injection site).
  Interventions: Drug: Kenalog

INTERVENTIONS:
Drug: Onabotulinumtoxin A — Intravaginal pelvic floor injection one series
  Other Names: Botox
  Arms: Onabotulinumtoxin A
Drug: Kenalog — Intravaginal pelvic floor injection one series
  Other Names: triamcinolone
  Arms: Kenalog

SUMMARY:
The goal of this study is to compare the effectiveness of two different medications used in intravaginal trigger point injections (injections into extremely painful areas of a muscle) to treat chronic pelvic pain. The study compares onabotulinumtoxinA (BOTOX®) (a drug prepared from the bacterial toxin botulin which temporarily paralyzes muscles) to Kenalog (a synthetic corticosteroid used as an anti-inflammatory agent).

DETAILED DESCRIPTION:
Chronic pelvic pain (CPP) is a common and often debilitating problem among women. The musculoskeletal system is an important factor in chronic pelvic pain. Studies have demonstrated that women with CPP had more frequent musculoskeletal findings. On physical examination, myofascial trigger points have been found. Trigger points are hyperirritable bands of muscle that can be felt from the vaginal wall. They are often knot-like or taut and are painful when pressure is placed on them. Intravaginal injections of these trigger points using steroids including Kenalog (triamcinolone) have been done and produced decreases in pelvic pain. Trigger point injections of Onabotulinumtoxin A has also been shown to decrease pain in subjects with CPP. This study will compare these two drugs and assess pain (using subject questionnaires) at one, three and six months post injection.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Healthy women > age 18 regardless of menopausal status
* Willing and able to fill out study questionnaires. In patients that are unable to read, the research nurse will be available to assist.
* High-tone pelvic floor dysfunction on vaginal exam
* A pelvic pain score of > 4 on screening Visual Analog Scale (VAS)
* Pain perceived to be in the pelvis that has been present for at least 3 months.

Exclusion Criteria:

* Patients that have had Botox to the bladder within the last 8 months
* Patients that have had Botox outside the bladder of > 160 u within the last 12 weeks.
* Patients that have had transvaginal trigger point injections of any form (Botox or steroid) in the last 3 months
* Pregnancy
* Concomitant use of any narcotic drug, alcohol, or any illicit drug use during the study period that could be deemed unsafe in combination with study medication as judged by the investigators.
* Any evidence of vaginitis on wet mount slide at initial visit that is untreated.
* Subject with any other vaginal epithelial disorder that could affect absorption of medication as deemed by the investigators.
* Any indication/condition/medication that the investigators identify as contraindicated in conjunction with study medication.
* Systolic blood pressure > 160 mm Hg on screening blood pressure
* Heart rate > 110 beats/minute on screening heart rate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03-26 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Bartley, DO, Principal Investigator — Beaumont
Locations (1):
- Beaumont Hospitals, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Onabotulinumtoxin A: Intervention is a one time 30 cc intravaginal injection totaling a dose of 200u of onabotulinumtoxin A and saline injected throughout the pelvic floor at 1, 3, 5, 7, 9 and 11 o'clock sites/locations.
  An injection of 30 cc of ropivicaine (5cc/6 sites) will be used, followed by a mixture of 200 u of Onabotulinumtoxin A and 6 cc of saline (1cc/injection site).
  Onabotulinumtoxin A: Intravaginal pelvic floor injection one series
- Kenalog: Intervention is a one time 30 cc intravaginal injection totaling a dose of 40mg/cc of Kenalog (triamcinolone) and ropivicaine 0.5% (29cc) injected throughout the pelvic floor at 1, 3, 5, 7, 9 and 11 o'clock sites/locations.
  A mixture of 40mg/1 cc of triamcinolone (40 mg) and 29cc of ropivicaine 0.5% (5cc/6 sites) will be used, followed by 6 cc of saline (1cc/injection site).
  Kenalog: Intravaginal pelvic floor injection one series
Period: 1 Month
Arm/Group | Onabotulinumtoxin A | Kenalog
Started | 10 | 11
Completed | 9 | 10
Not Completed | 1 | 1
Period: 3 Months
Arm/Group | Onabotulinumtoxin A | Kenalog
Started | 9 | 10
Completed | 9 | 8
Not Completed | 0 | 2
Period: 6 Months
Arm/Group | Onabotulinumtoxin A | Kenalog
Started | 9 | 8
Completed | 9 | 7
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Onabotulinumtoxin A | Kenalog | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.3) | 46.0 (12.8) | 46.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Pain Severity [Mean (Standard Deviation); unit: units on a scale] — Pain severity was constructed by averaging questions 3,4,5 and 6 of the Brief Pain Inventory (BPI) questionnaire (adding scores together and dividing by 4). Each question is on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). Thus, lower numbers represent a better outcome.
  units on a scale | 5.0 (1.7) | 4.9 (1.2) | 4.9 (1.4)
Pain Interference [Mean (Standard Deviation); unit: units on a scale] — The Pain Interference score was constructed by averaging the individual interference question scores from the BPI questionnaire (scores for questions 9A-9G added together and divided by 7). The questions assess how, during the past 24 hours, pain has interfered with general anxiety (9A), mood (9B), walking ability (9C), normal work (9D), relations with other people (9E), sleep (9F), and enjoyment of life (9G). Each question is scored on a scale from 0 (does not interfere) to 10 (completely interferes). Thus, a lower value represents a better outcome.
  units on a scale | 5.9 (2.3) | 4.7 (2.0) | 5.3 (2.2)
Pain Visual Analog Scale (VAS) [Median (Full Range); unit: units on a scale] — The pain visual analog scale (VAS) is a tool used by the patient to describe the intensity of their pain. Utilizing the visual analog scale, the patient describes their pain at baseline, before receiving trigger point injections. The visual analog scale ranges from 0 (no pain) to 10 (worst possible pain). Thus, a lower value represents a better outcome.
  units on a scale | 6 [5 to 8] | 5 [4 to 7] | 6 [4 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed by Change in Overall Pain Score Using the Visual Analog Scale (VAS).
Description: The visual analog scale asks subjects to rate their level of pain on a scale from 0-10, with 0 being 'No pain' and 10 being 'Worst pain imaginable', hence lower scores are better. The baseline and follow-up visual analog scale for pain was obtained at every visit regardless if the patient received Trigger Point Injections. The difference between visual analog scale at 1 month and the visual analog scale at baseline was calculated. Positive numbers indicate the pain increased from baseline to 1 month and negative numbers indicates that pain decreased.
Time Frame: Baseline and One Month
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 10
units on a scale | -2 [-4 to 0] | -1 [-2 to 3]
Statistical Analysis 1: Comparison: Onabotulinumtoxin A vs Kenalog; The null hypothesis assumed there were no differences in the pain score change between groups. Significance level was set at 0.05; Test type: Other; p = 0.072, Kruskal-Wallis; This test was selected since the distribution of the change in pain was not normal nor approximately symmetric

2. Primary Outcome: Pain Severity Assessed by Change in Overall Pain and Other Related Scores Using Questions 3, 4, 5, and 6 in the Brief Pain Inventory (BPI) Questionnaire.
Description: Pain severity was constructed by averaging questions 3,4,5 and 6 of the brief pain inventory questionnaire (adding scores together and dividing by 4). Each question is on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). Thus, lower numbers represent a better outcome. The difference between pain severity at 1 month and the pain severity at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 1 month and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and One Month
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 10
units on a scale | -0.03 [-1.75 to 3.25] | -0.88 [-1.25 to 2.0]
Statistical Analysis 1: Comparison: Onabotulinumtoxin A; The null hypothesis assumed there were no differences in the median change pain severity between the groups. Significance level was set at 0.05; Test type: Other; p = 0.624, Kruskal-Wallis

3. Primary Outcome: Pain Interference Assessed by Change in Overall Pain and Other Related Scores Using Questions 9A Through 9G in the Brief Pain Inventory (BPI) Questionnaire.
Description: The Pain Interference score was constructed by averaging the individual interference question scores from the brief pain inventory questionnaire (adding scores from questions 9A-9G and dividing by 7). The questions assess how, during the past 24 hours, pain has interfered with general anxiety (9A), mood (9B), walking ability (9C), normal work (9D), relations with other people (9E), sleep (9F), and enjoyment of life (9G). Each question is scored on a scale from 0 (does not interfere) to 10 (completely interferes). Thus, a lower value represents a better outcome. The difference between pain interference at 1 month and the pain interference at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 1 month and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and One Month
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 10
units on a scale | -0.14 [-4.71 to 3.57] | -0.36 [-1.86 to 2.29]
Statistical Analysis 1: Comparison: Onabotulinumtoxin A; The null hypothesis assumed that there is no difference in the change in pain interference between the groups. Statistical significance was set at 0.05; Test type: Other; p = 0.571, Kruskal-Wallis

4. Primary Outcome: Pain Assessed by Change in Overall Pain Symptom Using Question 2 of the Global Response Assessment (GRA) Questionnaire.
Description: The GRA questionnaire asks subjects to rate symptoms and functioning since having the research procedure, Trigger Point Injections (TPI). Question 2 asks the subject to rate their pain symptoms since having TPI. Scores are on a Likert scale, ranging from 1 (Markedly Worse) to 7 (Markedly Improved).
Time Frame: Baseline and One Month
Measure: Count of Participants; unit: Participants
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 10
Participants
  Markedly worse | 0 | 0
  Moderately worse | 1 | 0
  Mildly worse | 0 | 0
  Same | 2 | 5
  Slightly improved | 2 | 4
  Moderately improved | 3 | 1
  Markedly improved | 1 | 0
Statistical Analysis 1: Comparison: Onabotulinumtoxin A vs Kenalog; The null hypothesis assumed that there was no difference in the distribution between the groups. Significance level was set at 0.05; Test type: Other; p = 0.285, Kruskal-Wallis

5. Secondary Outcome: Pain Assessed by Change in Overall Pain Score Using the Visual Analog Scale (VAS) Questionnaire.
Description: The visual analog scale asks subjects to rate their level of pain on a scale from 0-10, with 0 being 'No pain' and 10 being 'Worst pain imaginable', hence lower scores are better. The baseline and follow-up visual analog scale for pain was obtained at every visit regardless if the patient received Trigger Point Injections. The difference between visual analog scale at 3 months and the visual analog scale at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 3 months and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and Three Months
Population: At 3 months, 9 subjects in the Onabotulinumtoxin A group completed the study and 8 completed in the Kenalog group. One subject in the Onabotulinumtoxin A did not have the pain assessed using the visual analog scale (missing data for this outcome, analysis conducted on 8 patients).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 8 | 8
units on a scale | -1 [-4 to 0] | -1 [-2 to 1]

6. Secondary Outcome: Pain Severity Assessed by Change in Overall Pain and Other Related Scores Using Questions 3, 4, 5, and 6 in the Brief Pain Inventory (BPI) Questionnaire.
Description: Pain severity was constructed by averaging questions 3,4,5 and 6 of the brief pain inventory questionnaire (adding scores and dividing by 4). Each question is on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). Thus, lower numbers represent a better outcome. The difference between pain severity at 3 months and the pain severity at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 3 months and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and Three Months
Population: At 3 months, 9 subjects in the Onabotulinumtoxin A group completed the study and 8 completed in the Kenalog group. One subject in the Onabotulinumtoxin A did not have information for pain severity (missing data for this outcome, analysis conducted on 8 patients).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 8 | 8
units on a scale | 0.25 [-1.75 to 2.75] | -0.37 [-2.75 to 3.25]

7. Secondary Outcome: Pain Interference Assessed by Change in Overall Pain and Other Related Scores Using Questions 9A Through 9G in the Brief Pain Inventory (BPI) Questionnaire.
Description: The Pain Interference score was constructed by averaging the individual interference question scores from the brief pain inventory questionnaire (adding scores together for questions 9A-9G and dividing by 7). The questions assess how, during the past 24 hours, pain has interfered with general anxiety (9A), mood (9B), walking ability (9C), normal work (9D), relations with other people (9E), sleep (9F), and enjoyment of life (9G). Each question is scored on a scale from 0 (does not interfere) to 10 (completely interferes). Thus, a lower value represents a better outcome. The difference between pain interference at 3 months and the pain interference at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 3 months and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and Three months
Population: At 3 months, 9 subjects in the Onabotulinumtoxin A group completed the study and 8 completed in the Kenalog group. One subject in the Onabotulinumtoxin A did not have information for pain interference (missing data for this outcome, analysis conducted on 8 patients).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 8 | 8
units on a scale | -0.21 [-2.71 to 2.0] | -1.0 [-3.71 to 3.71]

8. Secondary Outcome: Pain Assessed by Change in Overall Pain Symptom Using Question 2 of the Global Response Assessment (GRA) Questionnaire.
Description: as for outcome 4
Time Frame: Baseline and Three Months
Population: At 3 months, 9 subjects in the Onabotulinumtoxin A group completed the study and 8 completed in the Kenalog group. One subject in the Onabotulinumtoxin A did not have information for pain symptoms using question 2 in the global response assessment (missing data for this outcome, analysis conducted on 8 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 8 | 8
Participants
  Markedly worse | 0 | 0
  Moderately worse | 0 | 0
  Mildly worse | 1 | 1
  Same | 1 | 2
  Slightly improved | 1 | 3
  Moderately improved | 4 | 1
  Markedly improved | 1 | 1

9. Secondary Outcome: Pain Assessed by Change in Overall Pain Score Using the Visual Analog Scale (VAS) Questionnaire.
Description: The pain visual analog scale (VAS) is a tool used by the patient to describe their pain intensity. Utilizing the VAS, the patient describes their pain at baseline, before receiving trigger point injections. The VAS ranges from 0 (no pain) to 10 (worst possible pain). Thus, a lower value represents a better outcome.
Time Frame: Baseline and Six Months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 7
units on a scale | -1 [-6 to 2] | -1 [-5 to 2]

10. Secondary Outcome: Pain Severity Assessed by Change in Overall Pain and Other Related Scores Using Questions 3, 4, 5, and 6 in the Brief Pain Inventory (BPI) Questionnaire.
Description: Pain severity was constructed by averaging questions 3,4,5 and 6 of the brief pain inventory questionnaire (adding scores together and dividing by 4). Each question is on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). Thus, lower numbers represent a better outcome. The difference between pain severity at 6 months and the pain severity at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 6 months and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and Six Months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 7
units on a scale | 0.0 [-1.75 to 4.0] | -1.25 [-1.75 to 2.75]

11. Secondary Outcome: Pain Interference Assessed by Change in Overall Pain and Other Related Scores Using Questions 9A Through 9G in the Brief Pain Inventory (BPI) Questionnaire.
Description: The Pain Interference score was constructed by averaging the individual interference question scores from the brief pain inventory questionnaire (adding together scores for questions 9A-9G and dividing by 7). The questions assess how, during the past 24 hours, pain has interfered with general anxiety (9A), mood (9B), walking ability (9C), normal work (9D), relations with other people (9E), sleep (9F), and enjoyment of life (9G). Each question is scored on a scale from 0 (does not interfere) to 10 (completely interferes). Thus, a lower value represents a better outcome. The difference between pain interference at 6 months and the pain interference at baseline was calculated. Positive numbers indicate the pain severity increased from baseline to 6 months and negative numbers indicates that the severity of the pain decreased.
Time Frame: Baseline and Six months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 7
units on a scale | -0.71 [-1.71 to 4.0] | -1.14 [-5.0 to 2.43]

12. Secondary Outcome: Pain Assessed by Change in Overall Pain and Other Related Scores Using the Global Response Assessment (GRA) Questionnaire.
Description: The GRA questionnaire asks subjects to rate symptoms and functioning since having the research procedure, Trigger Point Injections (TPI). Scores are on a Likert scale, ranging from 1 (Markedly Worse) to 7 (Markedly Improved).
Time Frame: Baseline and Six Months
Measure: Count of Participants; unit: Participants
Arm/Group | Onabotulinumtoxin A | Kenalog
Number analyzed (Participants) | 9 | 7
Participants
  Markedly worse | 0 | 0
  Moderately worse | 1 | 0
  Mildly worse | 0 | 0
  Same | 2 | 2
  Slightly improved | 2 | 2
  Moderately improved | 2 | 3
  Markedly improved | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a 6 month period of time. Collection started at the initial trigger point injection visit and continued through the 6 month post-injection visit.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information does not differ from the clinicaltrials.gov definition. Adverse event collection was primarily collected by patient self-report. Additionally, the electronic medical record was reviewed at each visit, labs were evaluated and the physician researcher assessed the patient for adverse events as well.
Arm/Group | Onabotulinumtoxin A | Kenalog
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 5/10 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Onabotulinumtoxin A (N=10) | Kenalog (N=11)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 2 (3) | 0 (0)
Vaginal Yeast Infection (Renal and urinary disorders) | 2 (3) | 1 (1)
Increased Pelvic Pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Lower Extremity Numbness/Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Rib Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Exacerbation of Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute Kidney Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Rectal Spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Facial Abrasions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1)
Fecal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericoronitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT02369068/Prot_000.pdf
  • Informed Consent Form (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT02369068/ICF_001.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT02369068/SAP_002.pdf